CLINICAL TRIAL: NCT03359902
Title: Treatment of Mild Cognitive Impairment With Transcutaneous Vagal Nerve Stimulation
Acronym: TVNS MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201600730 -N-A; R21AG054876 (NIH); PRO00011145 (Other: UFIRST)
Record Dates: First submitted 2017-11-17; First posted 2017-12-02 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Vagal Nerve Stimulation; tVNS; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to either transcutaneous vagal nerve stimulation or sham for the first session, then switch to the other condition for their second session after a 1 week washout period.
Who Masked: Participant, Investigator
Masking Description: The sham stimulation experience is very similar to the tVNS stimulation experience. The electrodes are placed in a proximal location. Thus, without knowledge of the anatomy, the participants will be unable to determine which stimulation session is the tVNS one.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Initial tVNS (Experimental): This group will receive transcutaneous vagal nerve stimulation, initially. Participants will be randomized between the two arms of the crossover sessions (initial tVNS vs. initial Sham). Behavioral portions of the testing will then be carried out twice, with at least 72 hours between sessions (to avoid carryover effects).
  Interventions: Device: Transcutaneous vagal nerve stimulation; Device: Sham stimulation
- Initial Sham (Experimental): This group will receive sham stimulation, initially. Participants will be randomized between the two arms of the crossover sessions (initial tVNS vs. initial Sham). Behavioral portions of the testing will then be carried out twice, with at least 72 hours between sessions (to avoid carryover effects).
  Interventions: Device: Transcutaneous vagal nerve stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — Non-invasive stimulation provided by transcutaneous electrical nerve stimulation device at 20Hz, 100 μs pulse width
Device: Sham stimulation — Sham stimulation will be performed using electrodes placed on earlobe

SUMMARY:
Patients with amnestic mild cognitive impairment (MCI) often have compromised quality of life (QOL). Cognitive impairment is a major contributor to decrements in QOL and progression of MCI often leads to loss of independence and withdrawal from social participation. MCI, in many patients, is an early expression of neurodegenerative disease. Patients with MCI frequently convert to Alzheimer's disease (AD) (12-16 percent by some estimates per year). Treatments for MCI are of limited scope and availability and of limited effectiveness. Thus, there is great need for treatments that can improve cognition and extend QOL in patients with MCI. The investigators propose to investigate the effect of a non-invasive and safe intervention that should have direct influence on brain systems underlying AD, transcutaneous vagal nerve stimulation (tVNS).

DETAILED DESCRIPTION:
Patients with amnestic mild cognitive impairment (MCI) often have compromised quality of life (QOL). Cognitive impairment is a major contributor to decrements in QOL and progression of MCI often leads to loss of independence and withdrawal from social participation. MCI, in many patients, is an early expression of neurodegenerative disease. Patients with MCI frequently convert to Alzheimer's disease (AD) (12-16 percent by some estimates per year). Treatments for MCI are of limited scope and availability and of limited effectiveness. Thus, there is great need for treatments that can improve cognition and extend QOL in patients with MCI. The investigators propose to investigate the effect of a non-invasive and safe intervention that should have direct influence on brain systems underlying AD, transcutaneous vagal nerve stimulation (tVNS). Transcutaneous vagal nerve stimulation (tVNS) may ameliorate symptoms of MCI. The investigators have demonstrated, in patients with epilepsy, that VNS improves memory; however, tVNS has not been used to treat patients with MCI. tVNS can now be performed without surgery by transcutaneous stimulation of the auricular branch with electrodes on the external ear. tVNS has the potential to improve cognition and may even alter the course of decline in patients with MCI. The investigators will employ a multimodal MRI-based neuroimaging approach combined with comprehensive and targeted cognitive testing to assess changes with tVNS in cognition in patients with MCI.

The investigators will evaluate the effects of tVNS on patients who have been diagnosed with MCI as well as healthy older controls. Very little in the way of mechanistic data or understanding of individual differences in response to tVNS in MCI/AD has been published. Thus, this is a necessary study to evaluate the potential utility of tVNS to enhance cognitive performance in patients with MCI. These data may serve as a platform for supporting the development of a clinical treatment trial with this technology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with amnestic mild cognitive impairment/mild Alzheimer's disease
* Preservation of independence in functional abilities
* Healthy aged adults without MCI to serve as control group

Exclusion Criteria:

* Other medical or neurological conditions that may be associated with significant impaired cognition (e..g, moderate to severe traumatic brain injury, epilepsy, etc...)
* Vascular dementia or other non-AD spectrum diagnosed neurodegenerative disorders
* Significant current depression
* Uncorrected vision/hearing loss
* Unable to undergo MRI exam

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Williamson, Ph.D, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - McKnight Brain Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham First, Then tVNS: This group will receive sham stimulation, initially. Participants will be randomized between the two arms of the crossover sessions (tVNS first, then sham vs. sham first, then tVNS). Behavioral portions of the testing will then be carried out twice, with at least 72 hours between sessions (to avoid carryover effects).
  Transcutaneous vagal nerve stimulation: Non-invasive stimulation provided by transcutaneous electrical nerve stimulation device at 20Hz, 100 μs pulse width
  Sham stimulation: Sham stimulation will be performed using electrodes placed on earlobe
- tVNS First, Then Sham: This group will receive transcutaneous vagal nerve stimulation, initially. Participants will be randomized between the two arms of the crossover sessions (tVNS first, then sham vs. sham first, then tVNS). Behavioral portions of the testing will then be carried out twice, with at least 72 hours between sessions (to avoid carryover effects).
  Transcutaneous vagal nerve stimulation: Non-invasive stimulation provided by transcutaneous electrical nerve stimulation device at 20Hz, 100 μs pulse width
  Sham stimulation: Sham stimulation will be performed using electrodes placed on earlobe
Period: Overall Study
Arm/Group | Sham First, Then tVNS | tVNS First, Then Sham
Started | 41 | 18
Completed | 41 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Sham | Initial tVNS | Total
Number analyzed (Participants) | 41 | 18 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.56 (7.36) | 75.94 (6.96) | 75.81 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 20 | 4 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 39 | 17 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years of Education [Mean (Standard Deviation); unit: years] | 15.93 (2.78) | 16.44 (2.78) | 16.08 (2.77)
Wechsler Test of Adult Reading (standard score) [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Test of Adult Reading (WTAR) uses vocabulary level to estimate an individual's level of functioning before the onset of injury or illness. The raw score of the WTAR (0 worst, 50 best) is converted to a standard score (50-134), which is then used to predict full-scale IQ.
  units on a scale | 112.35 (12.11) | 110.89 (12.07) | 111.9 (12.01)
Beck Depression Inventory-2 [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-2 (BDI-II) is a 21-item self-report inventory measuring the severity of depression symptoms over the past two weeks. A total score of 0-9 indicates minimal symptoms,10-18 indicates mild symptoms, 19-29 indicates moderate symptoms, and 30-63 indicates severe symptoms.
  units on a scale | 8.32 (6.99) | 8.06 (6.32) | 8.24 (6.73)
Clinical Dementia Rating Scale (sum of boxes) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Dementia Rating (CDR) Scale is an assessment to stage severity of dementia. Cognitive functioning is rated on a 5 point scale (0 no impairment, 0.5 questionable impairment, 1 mild, 2 moderate, 3 severe) across 6 domains: memory, orientation, judgement & problem solving, community affairs, home & hobbies, and personal care. The CDR-some of boxes score (SOB) is obtained by summing each of the domain scores, with scores ranging from 0 to 18. Participants in the study must obtain a SOB of 0.5-4 to meet criteria for MCI diagnosis and qualify for the study.
  units on a scale | 0.66 (1.18) | 0.44 (0.16) | 0.59 (0.99)
Functional Activities Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The functional activities questionnaire (FAQ) is a 10-item screening tool for evaluating independence in instrumental activities for daily living. Sum of scores range 0 (fully independent) to 30 (fully dependent), and a cut-point of 9 is used to indicate impaired functioning.
  units on a scale | 3.27 (3) | 2.89 (2.74) | 3.15 (2.91)
Hopkins Verbal Learning Test (total immediate recall) [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Verbal Learning Test (HVLT-R) is a verbal learning and memory task with a 12-item word list learned over 3 trials. The total immediate recall score is the sum of correct words recalled after each of the 3 learning trials, which can range from 0 to 36.
  units on a scale | 17.46 (4.61) | 15.47 (3.94) | 16.88 (4.48)
Hopkins Verbal Learning Test (total delayed recall) [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Verbal Learning Test (HVLT-R) is a verbal learning and memory task with a 12-item word list learned over 3 trials. The total delayed recall score is the number of total correct words recalled (ranging from 0 to 12) after a 20-25 minute delay.
  units on a scale | 1.71 (2.44) | 1.94 (2.97) | 1.78 (2.58)
Hopkins Verbal Learning Test (total retention) [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Verbal Learning Test (HVLT-R) is a verbal learning and memory task with a 12-item word list learned over 3 trials. The total retention score is calculated by dividing the total delayed recall score by the higher score of learning trial 2 or 3, and multiplying this by 100, to provide the percentage of words retained following the 20-25 minute delay.
  units on a scale | 22.62 (30.03) | 26.67 (40.44) | 23.81 (33.10)
Hopkins Verbal Learning Test (recognition) [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Verbal Learning Test (HVLT-R) is a verbal learning and memory task with a 12-item word list learned over 3 trials. Within the delayed yes-no recognition part of the task, the participant is presented with a larger list or words and responds to whether each was on the original 12-item list. The recognition discrimination index score is calculated as number of hits (correctly identified words from the list) - number of false positive words (incorrectly identified words that were not on the list), with scores ranging from 0 to 12 (perfect score).
  units on a scale | 7.37 (2.67) | 7.35 (3.41) | 7.36 (2.88)

OUTCOME MEASURES:

1. Primary Outcome: Rey Auditory Verbal Learning Test (Total Delayed Recall)
Description: The Rey Auditory Verbal Learning Test (RAVLT) is a verbal learning and memory task with a 15-item word list learned over 5 trials. The total delayed recall score is the number of total correct words recalled (ranging from 0 to 15) after a 30 minute delay.
Time Frame: 30 minutes after administration of 5 list learning trials; 2 minutes to complete delayed recall of word-list
Population: As a crossover design, each participant operated as their own control. Therefore results of data analysis are presented per intervention (i.e., tVNS vs. Sham) rather than per arm (i.e., first tVNS, then Sham, etc.).
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Sham: This is the sham arm for all participants.
  Sham stimulation: Sham stimulation will be performed using electrodes placed on earlobe
- tVNS: This is the active stimulation arm of all participants.
  Behavioral portions of the testing will then be carried out twice, with at least 72 hours between sessions (to avoid carryover effects).
  Transcutaneous vagal nerve stimulation: Non-invasive stimulation provided by transcutaneous electrical nerve stimulation device at 20Hz, 100 μs pulse width
Arm/Group | Sham | tVNS
Number analyzed (Participants) | 58 | 58
score on a scale | 6.43 [0 to 15] | 7.83 [0 to 15]
Statistical Analysis 1: Comparison: Sham vs tVNS; A linear mixed effects model was conducted to account for carryover and order effects in this crossover trial. Assuming α = 0.05, two-sided test, and 60 participants in total. If the carryover effect is negligible, we will have 90% power to detect an effect size of 0.604 for memory improvement; Test type: Superiority; p = 0.11, Mixed Models Analysis; beta = 1.4

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 month.
Arm/Group | Initial Sham | Initial tVNS
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT03359902/Prot_003.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03359902/SAP_004.pdf
  • Informed Consent Form (2021-09-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03359902/ICF_002.pdf